CLINICAL TRIAL: NCT02037347
Title: Palifermin Treatment of Toxic Epidermal Necrolysis
Brief Title: Study to Evaluate the Use of Palifermin to Treat Toxic Epidermal Necrolysis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment numbers precluded completion of the study during a reasonable amount of time.
Sponsor: Brett King (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor-Investigator, Brett King, Assistant Professor of Dermatology, Yale University
Organization: Yale University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0901004673; 020901 (Other: Bridgeport Hospital)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Toxic Epidermal Necrolysis; Stevens-Johnson Syndrome
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palifermin (Experimental): Palifermin 60 micrograms/kg/day IV for 3 consecutive days
  Interventions: Drug: Palifermin

INTERVENTIONS:
Drug: Palifermin
  Other Names: Kepivance

SUMMARY:
To test the ability of palifermin (a recombinant human keratinocyte growth factor) to decrease mucocutaneous injury and to promote epithelial repair in Toxic Epidermal Necrolysis and Stevens-Johnson Syndrome-Toxic Epidermal Necrolysis Overlap, diseases in which there is extensive sloughing of the skin and mucosa, including that of the eyes, gastrointestinal tract, respiratory and genitourinary systems.

ELIGIBILITY:
Inclusion Criteria:

* Skin biopsy in early disease showing apoptotic keratinocytes in the epidermis and in more advanced disease necrosis of the entire epidermis
* Epidermal detachment or erythematous to purpuric macules involving more than 10% of body surface area in addition to involvement of the oropharynx; there may be further involvement of other mucosal surfaces, ie. conjunctivae, gastrointestinal tract, respiratory and genitourinary epithelia
* Age of 18 years old or older
* The patient is expected to survive longer than 48 hours

Exclusion Criteria:

* Skin detachment above 90% of the body surface area
* Skin detachment has not progressed during the previous 48 hours
* A positive serum pregnancy test
* Age < 18 years old
* Known hematologic or solid organ malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale-New Haven Hospital, New Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palifermin
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 73-year-old male.
Arm/Group | Palifermin
Number analyzed (Participants) | 1
Age, Customized [Number; unit: years]
  Age | 73
Sex/Gender, Customized [Number; unit: participants]
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Time-to-cutaneous Re-epithelialization
Time Frame: The number of days between the start of palifermin administration and complete re-epithelialization of skin up to 14 days
Measure: Number; unit: days
Arm/Group | Palifermin
Number analyzed (Participants) | 1
days | 6

2. Secondary Outcome: Time-to-mucosal Re-epithelialization
Time Frame: The number of days between the start of palifermin administration and complete re-epithelialization of oral mucosa up to 14 days
Population: Adverse event experienced by participant precluded measuring this outcome.
Arm/Group | Palifermin
Number analyzed (Participants) | 0

3. Secondary Outcome: Time-to-cessation of Epidermal Necrosis
Time Frame: The number of days between the start of palifermin administration and cessation of further epidermal necrosis up to 14 days
Measure: Number; unit: days
Arm/Group | Palifermin
Number analyzed (Participants) | 1
days | 3

ADVERSE EVENTS:
Arm/Group | Palifermin
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin (N=1)
ischemic necrosis (Gastrointestinal disorders) | 1 — ischemic necrosis of the small bowel

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes